CLINICAL TRIAL: NCT02424747
Title: Long Term Survival and Renal Outcomes in Critically Ill Patients After Acute Kidney Injury: Swedish Multi-centre Cohort Study
Brief Title: Long-term Survival and Renal Outcomes in Critically Ill Patients After Acute Kidney Injury: Swedish Multi-centre Cohort Study
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Claire Rimes-Stigare, MD, Karolinska Institutet
Other Study IDs: Karolinska Institutet SIR
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- De Novo Acute Kidney Injury: Patients who developed Acute Kidney Injury during intensive care admission and not previously diagnosed with chronic kidney disease or end stage renal disease.
  Interventions: Other: Acute Kidney Injury
- No Acute Kidney Injury.: Intensive care patients not diagnosed with acute kidney Injury during admission and not previously diagnosed with Chronic Kidney Disease or End Stage Renal Disease.

INTERVENTIONS:
Other: Acute Kidney Injury — We will identify and observe "exposure" to Acute Kidney Injury during Intensive Care admission.
  Groups: De Novo Acute Kidney Injury

SUMMARY:
The study evaluates how outcome varies among critically ill patients with and without acute kidney injury. Data from the Swedish Intensive care register and other Swedish national registers is used to compare how survival and post discharge renal function differ between critically ill patients with and without acute kidney injury.

DETAILED DESCRIPTION:
Background: Acute kidney injury is common amongst intensive care patients and is associated with extremely high mortality and morbidity in terms of increased risk of developing Chronic Kidney Disease (CKD) and End Stage Renal Disease (ESRD). Patients with CKD are at increased risk of cardiovascular, cerebro-vascular disease and long term increased risk of death. Those patients who progress to ESRD have a 20% mortality risk per year in Sweden. Outcome after acute kidney injury in the Swedish critical care population has never previously been described.

Method: This cohort study uses Swedish national healthcare registers to investigate the epidemiology of acute kidney injury. The Swedish Intensive Care Register (SIR) provides the population base, with data extraction between 2005 and 2011. The information obtained is cross-matched by the Swedish board for health and welfare (Social Styrelsen) with other national registries. All data are returned anonymized and individual patients can not be identified in any way. Additionally analysis is performed on a group and not on an individual basis. The key to this data is held by Swedish board for health and welfare. The other national registries include the Swedish Cause of Death Register (Dödsregister), the Swedish renal register (Svensknjurregistret) and the in and out-patients registers (Öppen- slutenvårdsregister) these are used to obtain data on all cause mortality, co-morbidities, Pre and Post ICU CKD and ESRD. Epidemiological methods are used to analyse the data.

Investigators aim to describe outcome in terms of long-term mortality (up to five years) and renal morbidity (incidence of CKD and ESRD) in critically ill patients with and without de novo AKI in Sweden.

ELIGIBILITY:
Inclusion Criteria:

All first admissions of adult patients registered on the Swedish Intensive Care Register between January 1st 2005 and January 1st 2011.

Exclusion Criteria:

Patients under 18. Subjects with incomplete records. Patients previously diagnosed with Chronic Kidney Disease or End Stage Renal disease.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was provided by the Swedish Intensive Care register and included patients receiving intensive care treatment between January 2005 and January 2011
Sampling Method: Non-Probability Sample
Enrollment: 103000 (Actual)
Dates: Start 2005-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 5 year

SECONDARY OUTCOMES:
Incidence of Chronic Kidney Disease | 5 years
Incidence of End Stage Renal Failure | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Claire Stigare, MD, Principal Investigator — karolinska University Hospital, Karolinska Institute

REFERENCES:
- [Background] Goldstein SL, Jaber BL, Faubel S, Chawla LS; Acute Kidney Injury Advisory Group of American Society of Nephrology. AKI transition of care: a potential opportunity to detect and prevent CKD. Clin J Am Soc Nephrol. 2013 Mar;8(3):476-83. doi: 10.2215/CJN.12101112. PMID 23471414
- [Background] Bellomo R. The epidemiology of acute renal failure: 1975 versus 2005. Curr Opin Crit Care. 2006 Dec;12(6):557-60. doi: 10.1097/01.ccx.0000247443.86628.68. PMID 17077686
- [Background] Rimes-Stigare C, Awad A, Martensson J, Martling CR, Bell M. Long-term outcome after acute renal replacement therapy: a narrative review. Acta Anaesthesiol Scand. 2012 Feb;56(2):138-46. doi: 10.1111/j.1399-6576.2011.02567.x. Epub 2011 Oct 19. PMID 22092145
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] Bellomo R, Kellum JA, Ronco C. Acute kidney injury. Lancet. 2012 Aug 25;380(9843):756-66. doi: 10.1016/S0140-6736(11)61454-2. Epub 2012 May 21. PMID 22617274
- [Background] Emilsson L, Lindahl B, Koster M, Lambe M, Ludvigsson JF. Review of 103 Swedish Healthcare Quality Registries. J Intern Med. 2015 Jan;277(1):94-136. doi: 10.1111/joim.12303. Epub 2014 Sep 27. PMID 25174800
- [Background] Adami HO, Hernan MA. Learning how to improve healthcare delivery: the Swedish Quality Registers. J Intern Med. 2015 Jan;277(1):87-9. doi: 10.1111/joim.12315. Epub 2014 Nov 24. No abstract available. PMID 25270255
- [Derived] Rimes-Stigare C, Frumento P, Bottai M, Martensson J, Martling CR, Bell M. Long-term mortality and risk factors for development of end-stage renal disease in critically ill patients with and without chronic kidney disease. Crit Care. 2015 Nov 3;19:383. doi: 10.1186/s13054-015-1101-8. PMID 26526622